CLINICAL TRIAL: NCT01415024
Title: Resynchronization in Paced Heart Failure Patients With ICD Indication
Brief Title: Resynchronization in Paced Heart Failure Patients With Implantable Cardioverter Defibrillator (ICD) Indication
Acronym: CRTICD Dual LV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Schuechtermann-Klinik (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Dr. med. Wolfgang Kranig, Schuechtermann- Klinik
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BO/01/2011
Record Dates: First submitted 2011-07-28; First posted 2011-08-11 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Heart Failure; Left Bundle-Branch Block
Keywords: CRT; Dual LV; Triple Ventricle stimulation; two leftventricular leads; Av VV optimization; Lv dp/dt measurement
MeSH Terms: conditions — Heart Failure; Bundle-Branch Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: second LV lead in CRT — second LV lead in CRT

SUMMARY:
Today patients with a Cardiac Resynchronization Therapy (CRT) indication usually receive 2 ventricular leads, right ventricular (RV) apex and left ventricular (LV) (postero-) lateral, gaining a responder rate of approximately 70%. However, the physiological agitation of the left ventricle takes place over two pathways. Therefore single point stimulation might be insufficient for a dilated, insufficiently and asynchronously contracting left ventricle, resulting in either insufficient or no response to the therapy.

In the "CRT ICD Dual LV" study the patients receive a second LV lead in an anterior vein. When this lead is placed, temporary dual LV stimulation is started. To assess the effectivity of the dual LV lead stimulation intraoperatively a LV dp/dt-pressure measurement is taken. If there is an increase in LV dp/dt, the patients will be stimulated with both leads permanently. If not they will be stimulated conventionally.

The patients participating in this study are monitored for 12 months after implantation.

ELIGIBILITY:
Inclusion Criteria:

* EF less than 35 percent
* CAD or dilatative Cardiomyopathy
* Sinus rhythm
* NYHA III or IV, stable recompensated
* QRS more than 120ms
* LBBB
* Patient signed Consent Form
* Age more than 18 and less than 80 y

Exclusion Criteria:

* permanent atrial Fibrillation
* permanent AV-Block II or III
* Tricuspidal- and or artificial aortic valve
* Indication for ACB or ACB less than 3 months ago
* myocardial infarction less than 3 months
* hypertrophic obstructive Cardiomyopathy; constrictive Pericarditis
* heartfailure with iv catecholamine therapy
* Manifested, uncontrolled, Hypo- oder Hyperthyreosis
* Severe renal insufficiency with Creatinine more than 2,5 mg per dL
* patients, who did not sign the consent form
* General medical conditions, which restrict the patient compliance
* Participation in another study
* life expectancy less than 1 y
* Age less than 18 y or more than 80y
* Pregnant women or Women of childbearing age

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
LV dp/dt pressure during dual LV CRT stimulation vs. conventional biventricular pacing | Implantation with pressure measurement will take place in the first week

SECONDARY OUTCOMES:
Leftventricular endsystolic volume | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Kranig, MD, Principal Investigator — Schuechtermann-Klinik
Locations (1):
- Schuechtermann-Klinik, Bad Rothenfelde, Lower Saxony, Germany